CLINICAL TRIAL: NCT01525303
Title: Additive Effects of Aerobic Exercise to a Standard Behavioral Self-Management Program for Chronic Headaches
Brief Title: Effects of Aerobic Exercise Within a Behavioral Treatment Program for Chronic Headaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Donald Penzien, Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0044
Record Dates: First submitted 2012-01-30; First posted 2012-02-02 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Headaches
Keywords: headaches; behavioral treatment; physical activity
MeSH Terms: conditions — Headache Disorders; Headache; Motor Activity | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise-Start (ES) (Experimental): The ES group will receive standard behavioral treatment in the Self-Management Training Program for Chronic Headaches. In addition to this material, participants in this group will receive an exercise prescription for 20 minutes of moderate-intensity aerobic activity at the beginning of Week 1. The exercise prescription will increase to 25 minutes in Week 2, and 30 minutes in Week 3. They are asked to maintain 30 minutes per day of exercise through Week 8. Participants choose the type of exercise, and have the option to break it up into 10-minute increments throughout the day.
  Interventions: Behavioral: Behavioral Treatment for Chronic Headache- Exercise Version
- Exercise-Middle (EM) (Experimental): The EM group will receive standard behavioral treatment in the Self-Management Training Program for Chronic Headaches.In addition to this material, participants in this group will receive an exercise prescription for 20 minutes of moderate-intensity aerobic activity at the beginning of Week 5. The exercise prescription will increase to 25 minutes in Week 6, and 30 minutes in Week 7. They are asked to maintain 30 minutes per day of exercise through Week 8. Participants choose the type of exercise, and have the option to break it up into 10-minute increments throughout the day.
  Interventions: Behavioral: Behavioral Treatment for Chronic Headache- Exercise Version

INTERVENTIONS:
Behavioral: Behavioral Treatment for Chronic Headache- Exercise Version — This behavioral treatment program consists of behavioral approaches to headache management: progressive muscle relaxation, stress-management training, and biofeedback. Skills for these techniques are presented during the clinic sessions, and supplemented with workbooks and audio CDs. In addition, all participants will receive a graduated exercise prescription of 20-30 minutes of moderate-intensity exercise, five days per week. They will be instructed to assess the intensity of their exercise using the Borg perceived exertion scale. Client contact sessions are as follows: Clinic Session (CS)1; Phone Session (PS) 1 (end of week1), CS 2 (end of week 4); PS 2 (end of week 6); CS 3 (end of week 8).

SUMMARY:
This proposed study seeks to examine whether adding an aerobic exercise prescription to a behavioral treatment program for chronic headaches will improve headache frequency and intensity, headache-related disability, and mood. It is hypothesized that participants who receive the exercise prescription at the start of treatment will show greater gains than those who receive the prescription halfway through treatment. It is also predicted that participants who begin the exercise component halfway through treatment will demonstrate greater improvement in the second half of treatment compared to the first half.

DETAILED DESCRIPTION:
Aerobic exercise has long been discussed as a potential treatment for chronic headaches, though research in this area has been somewhat limited. It is warranted to consider the effectiveness of aerobic exercise as part of a larger headache management intervention. Early research in this area suggests that including an exercise component in conjunction with other effective forms of headache management, such as progressive muscle relaxation, biofeedback, and stress management, is associated with improvement in number of days with a headache, headache pain intensity and mood. None of these studies have specifically analyzed the effectiveness of the aerobic exercise component, though Lemestra et al. (2002) noted that participants who continued with their exercise regimen had better overall outcomes three months after the intervention ended.

Given the high rates of obesity and the fact that many people do not meet the minimum daily requirement for exercise, it is worthwhile to investigate the additive effect of exercise to behavioral headache interventions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic headache (according to International Headache Association (IHA) guidelines) by research personnel
* Interested in receiving behavioral treatment for chronic headaches
* Engaged in less than 60 minutes/week of physical activity in the past 3 months
* Physically capable of engaging in a regular exercise routine
* Interested in in taking part in a regular exercise routine
* Regular internet access (at least once a week)

Exclusion Criteria:

* Males
* Unable to access internet at least once a week
* Currently engaging in regular exercise
* Not interested in participating in regular exercise
* Not capable of safely exercising
* Pregnant, nursing, or planning on becoming pregnant during the course of the study
* Does not meet IHA diagnostic criteria for chronic headache
* Not interested in behavioral headache treatment
* Diagnosis of Medication Overuse Headache, or headaches related to a physical or neurological disorder
* Cognitive or other forms of impairment that would decrease ability to fully engage in treatment

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Patient-reported headache-free days per week | 2 weeks prior to treatment through 2 weeks post-treatment
  Patients are asked to report the number of days per week they do no experience headaches

SECONDARY OUTCOMES:
Headache Disability Index (HDI) | baseline, 8 weeks, 10 weeks
  HDI is a 25-item questionnaire that assesses headache-related functional and emotional disability in chronic headache sufferers. Participants respond to items using a 3-point scale: "yes," "sometimes," or "no."
Highest weekly headache intensity | 2 weeks prior to treatment through 2 weeks post-treatment
  Patients are asked to report the the intensity of their worst headache during the past week, using a 0 (pain-free) to 10 (extremely intense pain) scale.
Composite Depression/Anxiety Screening Scale (PHQ-4) | 2 weeks prior to treatment through 2 weeks follow-up
  This is a 4-item measure assessing symptoms of anxiety and depression in the past two weeks. Participants respond on a 4 point scale: 0=Not at all; 1=Several days; 2=More than half of the days; 3=Nearly every day. When this measure is administered during the course of treatment (weekly) participants will be asked to respond based on their experiences in the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Penzien, Ph.D., Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States